CLINICAL TRIAL: NCT01211743
Title: Study of Oxidative Stress in Standard Laparoscopic vs Single Port Cholecystectomy for Uncomplicated Cholelithiasis (Lap vs SILS)
Brief Title: Oxidative Stress in Standard Laparoscopic vs Single Port Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: G. Hatzikosta General Hospital (Other)
Collaborators: Demokrition University of Thrace (Other); University of Ioannina (Other)
Responsible Party: George Pappas-Gogos MD, G Hatzikosta General Hospital of Ioannina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GH-1948-06
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Uncomplicated Cholelithiasis; Cholecystectomy; Laparoscopy; Standard Technique; Single Port Laparoscopy
Keywords: SILS; Oxidative Stress; 8-epiPGF2a; SILS vs standard laparoscopic cholecystectomy
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lap Group (Active Comparator): Patients in this group are operated for uncomplicated cholelithiasis with standard 4 port laparoscopic cholecystectomy
  Interventions: Other: Laparoscopic cholecystectomy; Other: Single incision laparoscopic cholecystectomy
- SILS group (Active Comparator): Patients in this group are operated for uncomplicated cholelithiasis with Single Incision Laparoscopic Cholecystectomy
  Interventions: Other: Single incision laparoscopic cholecystectomy

INTERVENTIONS:
Other: Laparoscopic cholecystectomy — Standard 4 port laparoscopic cholecystectomy
  Arms: Lap Group
Other: Single incision laparoscopic cholecystectomy — One port placed through the umbilicus

SUMMARY:
Study of Oxidative Stress Markers in order to assess whether there are differences between standard laparoscopic cholecystectomy vs single port cholecystectomy for uncomplicated cholelithiasis

ELIGIBILITY:
Inclusion Criteria:Uncomplicated cholelithiasis American Society of Anesthesiologists (ASA) I or II No previous operations in upper abdomen Body mass index (BMI) -

Exclusion Criteria:Cholecystitis ASA > II BMI>30 Previous operations in upper abdomen Previous operations in intestine Smokers Alcohol Drugs

-

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- G Hatzikosta General Hospital of Ioannina, Ioannina, Epirus, Greece

REFERENCES:
- [Derived] Pappas-Gogos G, Tellis CC, Trypsianis G, Tsimogiannis KE, Tsimoyiannis EC, Simopoulos CE, Pitiakoudis M, Tselepis AD. Oxidative stress in multi-port and single-port cholecystectomy. J Surg Res. 2015 Mar;194(1):101-6. doi: 10.1016/j.jss.2014.09.020. Epub 2014 Sep 28. PMID 25438954